CLINICAL TRIAL: NCT05186129
Title: To Determine the Bioequivalence of Clopid® (Clopidogrel) 75 mg Tablet Manufactured by Ferozsons Laboratories Ltd. Pakistan and Plavix® 75 mg Tablet Manufactured by Sanofi Winthrop Industrie France for Sanofi Pakistan After Oral Administration to Healthy Adult Male Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Clopid® (Clopidogrel) 75 mg Tablet and Plavix® 75 mg Tablet After Oral Administration to Healthy Adult Subjects Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Center for Bioequivalence Studies and Clinical Research (Other)
Collaborators: Ferozsons Laboratories Ltd. (Industry)
Responsible Party: Principal Investigator, Dr. Naghma Hashmi, Sub Investigator, Center for Bioequivalence Studies and Clinical Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-024-CLO-2017/Protocol/1.0
Record Dates: First submitted 2021-12-16; First posted 2022-01-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Bioequivalence
Keywords: Clopidogrel; Platelet Aggregation Inhibitor; Bioequivalence
MeSH Terms: interventions — Tablets; Clopidogrel

STUDY DESIGN:
Intervention Model Description: open label, randomized, single-dose, 2 way cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clopid® 75 mg(Clopidogrel)Tablet of Ferozsons Laboratories Ltd. Pakistan (Experimental): Single dose of Clopid® 75 mg Tablet administered under fasting condition
  Interventions: Drug: Clopid® 75 mg Tablet
- Plavix® 75mg Tablet of Sanofi Winthrop Industrie France for Sanofi Pakistan. (Active Comparator): Single dose of Plavix® 75 mg Tablet administered under fasting condition
  Interventions: Drug: Plavix® 75mg Tablet

INTERVENTIONS:
Drug: Clopid® 75 mg Tablet — Single dose of Clopid® 75 mg Tablet (Clopidogrel) was administered after a 10-hour overnight fast.
  Other Names: Clopidogrel
  Arms: Clopid® 75 mg(Clopidogrel)Tablet of Ferozsons Laboratories Ltd. Pakistan
Drug: Plavix® 75mg Tablet — Single dose of Plavix® 75 mg Tablet (Clopidogrel) was administered after a 10-hour overnight fast.
  Other Names: Clopidogrel
  Arms: Plavix® 75mg Tablet of Sanofi Winthrop Industrie France for Sanofi Pakistan.

SUMMARY:
To compare the rate and extent of absorption of Clopid® (Clopidogrel) 75 mg Tablet and Plavix® (clopidogrel) 75 mg tablet under fasting condition.

DETAILED DESCRIPTION:
Single dose, Randomized, Open-label, 2-Way Crossover, Bioequivalence Study of Clopid® of Ferozsons Laboratories Limited and Plavix® of Sanofi Winthrop Industrie France for Sanofi Pakistan Following a 75 mg Dose In Healthy Subjects Under Fasting Condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects , age between 18 to 55 years old
* Body mass index (BMI) between 18.5-30.0 kg /m2.
* Subject is willing to participate and to Sign written informed consent form
* Subjects should have a blood pressure after resting for at least three minutes between 100-139 mmHg (systolic) and 60-89 mmHg (diastolic).
* Subjects should have a supine (ECG) heart rate between 60 and 100 beats/min after resting for at least 3 minutes.
* Ability to fast for 10 hours and consume standard meal.
* Subjects must be in good health as determined by medical history, physical exmination, ECG, vital signs, medical tests including biochemistry, urinalysis, serology and hematology in serum/urine.

Exclusion Criteria:

* • History of smoking , alcoholism, and a positive test for drugs of abuse, heavy pan or gutka user as judged by teeth / mouth inspection.

  * Subjects with clinically relevant evidence of cardiovascular, gastrointestinal/hepatic, renal, psychiatric, respiratory, urogenital, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery or other relevant diseases as revealed by medical history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constitute a risk factor when taking study medication.
  * Subjects allergic to Clopidogrel and/or, subjects who received any investigational drug within four weeks prior to screening.
  * Intake of Smokeless tobacco, Tea, Coffee or other xanthenes derivatives (e.g. chocolate, cocoa) and poppy seeds 48 hours prior to study Check- In and must not consume grape fruit or juice of grape fruit at least 14 days prior to study.
  * Donation or loss of more than 450 mL of blood within 3 months prior to the screening.
  * Ingestion of OTC drug, within 14 days of drug administration (e.g. aspirin, ibuprofen)
  * History of intake of any prescribed medicine during a period of 30 days, prior to drug administration day of study.
  * Other prescription medication such as Antidepressent (Bupripion), CYP2C19 inhibitors (cimetidine, esomeprazole, etravirine, felbamate, fluconazole, fluoxetine, fluvoxamine, ketoconazole, omeprazole, ticlopidine, voriconazole), Macrolide and related antibiotics (erythromycin, telithromycin), Proton pump inhibitors (esomeprazole, omeprazole), Rifamycins (rifampin) and Anti-Coagluant (Warfarin) should also not be taken before 14 days.
  * Individuals who had undergone any major surgery within 3 months prior to the start of the study, unless deemed eligible by the Principal Investigator or whomever he/she may designate.
  * Subject has a history of any illness that, in the opinion of investigator might confound the result of the study or post additional risk in administrating Clopidogrel to the subject.
  * Subjects having any external wound.
  * Inability to take oral medication.
  * Subjects with clinically significant abnormalities in investigations (safety assessments) as determined by the Investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male Pakistani subjects
Enrollment: 36 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-36 hours post dose
  maximum plasma concentration
AUC | 0-36 hours post dose
  Area under plasma concentration time curve

SECONDARY OUTCOMES:
Tmax | 0-36 hours post dose
  time to reach maximum plasma concentration
t 1/2 | 0-36 hours post dose
  Terminal half-life
Incidence of Treatment-Emergent Adverse Event | 0-36 hours post dose
  safety and tolerability of Experimental drug Clopid® (Clopidogrel) 75 mg Tablet and Comparator drug Plavix® 75mg Tablet in Pakistani population

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Muhammad R Raza, PhD, Principal Investigator — Center for Bioequivalence Studies and Clinical Research
Locations (1):
- Center for Bioequivalence Studies and Clinical Research (CBSCR) ICCBS, University of Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The study related information can be obtained via proper request to the Co-PI/PI unless the confidentiality of the participants are not compromised